CLINICAL TRIAL: NCT06306170
Title: Efficacy of Advanced Radiotherapy (ART) in Gynecological Cancer Patients (GYN-ART)
Brief Title: Advanced Radiotherapy (ART) in Gynecological Cancer Patients (GYN-ART)
Acronym: GYN-ART
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Andrei Fodor, MD, MD, IRCCS San Raffaele
Other Study IDs: GYN-ART
Record Dates: First submitted 2024-02-14; First posted 2024-03-12 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Gynecologic Cancer; Radiotherapy Side Effect; Radiotherapy; Complications; Survivorship; Progression, Disease; Progression, Clinical
Keywords: Gynecologic Cancer; Image Guided Radiotherapy; PET/CT; Intensity Modulated Radiotherapy; Stereotactic Body Radiotherapy; Oligometastases
MeSH Terms: conditions — Radiation Injuries; Disease Progression | interventions — Radiotherapy, Image-Guided; Radiotherapy, Intensity-Modulated; Radiosurgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gynecologic cancer patients: Gynecologic cancer patients treated with IGRT, IMRT, SBRT (advanced radiotherapy-ART)
  Interventions: Radiation: Image Guided Radiotherapy

INTERVENTIONS:
Radiation: Image Guided Radiotherapy — Patients treated with IGRT, IMRT, SBRT for Gynecological cancer will be evaluated
  Other Names: Intensity Modulated Radiotherapy; Stereotactic Body Radiotherapy

SUMMARY:
This is an observational mono-institutional study. Patients with gynecologic tumors treated with advanced radiotherapy- Image Guided Radiotherapy (IGRT), Intensity Modulated Radiotherapy (IMRT), Stereotactic Body Radiotherapy (SBRT)- will be included and toxicity and outcomes analyzed.

DETAILED DESCRIPTION:
The patients with gynecological cancer treated with Advanced Radiotherapy (ART)- Image Guided Radiotherapy (IGRT), Intensity Modulated Radiotherapy (IMRT), Stereotactic Body Radiotherapy (SBRT)- at the Department of Radiotherapy of "IRCCS San Raffaele Scientific Institute" (IRCCSSRaffaele) from January 2005 to January 2024 will be identified and their clinical and dosimetric data retrieved and analyzed.

The study objectives are the analysis of acute and late toxicity, and clinical outcomes, such as local, regional and distant control,disease free survival, cancer-specific survival, and overall survival. Secondary objective is the identification of prognostic factors for toxicity, disease progression, survival, including radiomic characteristics.

ELIGIBILITY:
Inclusion Criteria:

* gynecologic cancer patients
* >18 years old
* treated with advanced radiotherapy techniques (IGRT, IMRT, SBRT)

Exclusion Criteria:

* other tumors
* > 90 years old

Ages: 18 Years to 90 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Gynecologic tumor patients
Study Population: Gynecologic cancer patients, > 18 years old, treated with IGRT, IMRT, SBRT
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2027-02-15 (Estimated); Study Completion 2029-02-15 (Estimated)

PRIMARY OUTCOMES:
Local Relapse Free Survival | From date of radiotherapy end until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 120 months
  local control (on the treated site) of the disease
Regional Relapse Free Survival | From date of radiotherapy end until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 120 months
  regional control (regional lymph nodal chain) of the disease
Distant Metastases Free Survival | From date of radiotherapy end until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 120 months
  distant metastases developed after the treatment
Disease Free Survival | From date of radiotherapy end until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 120 months
  absence of disease progression during the follow-up
Overall Survival | From date of radiotherapy end until the date of death from any cause, assessed up to 120 months
  survival from all causes
Cancer Specific Survival | From date of radiotherapy end until the date of death from disease progression, assessed up to 120 months
  cancer survival

SECONDARY OUTCOMES:
Acute toxicity | Up to three months from the start of radiotherapy
  Toxicity developed in the first three months after the treatment, assessed with Common Terminology Criteria for Adverse Events (CTCAE) v5.0 scale, which displayes grades from 1 to 5, with grade 1 meaning mild toxicity and grade 5 death related to toxicity
Late toxicity | From three months after the start of radiotherapy until the end of follow-up or death, assessed up to 120 months
  Toxicity developed after three months until the end of follow-up or death, assessed with Common Terminology Criteria for Adverse Events (CTCAE) v5.0 scale, assessed with Common Terminology Criteria for Adverse Events (CTCAE) v5.0 scale, which displayes grades from 1 to 5, with grade 1 meaning mild toxicity and grade 5 death related to toxicity

OTHER OUTCOMES:
Predictive factors for disease progression and death | From radiotherapy end to date of local, regional progression, distant failure, or death, assessed up to 120 months
  Factors predicting survival. Survival trees, univariate/multivariate Cox regression models will be estimated to identify potential risk factors associated with survival outcomes
Radiomic predictive factors for disease progression and death | From radiotherapy end to the first registered event (disease progression or death), assessed up to 120 months
  CT and PET/CT radiomic features predicting relapse or death will be extracted, acording to IBSI (Image Biomarker Standardisation Initiative), owning to the different families of features: Morphology, Statistical, Intensity Histogram, Grey Level Cooccurrence Matrix 3D-average, Grey Level Co-occurrence Matrix 3D-combined, Grey Level Run Lenght 3D-average. Grey Level Run Lenght 3D_combined, Grey Level Size Zone Matrix 3D, Neighbors Grey Tone Difference Matrix 3D, Grey Level Distance Zone Matrix 3D, standard convolutional filters within radiomic workflow (wavelets, Laplacian of Gaussian)

CONTACTS AND LOCATIONS:
Overall Officials: andrei Fodor, MD, Principal Investigator — IRCCS San Raffaele Scientific Institute
Locations (1):
- San Raffaele Scientific Institute, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study (anonymized individual participant data) are available on request from the corresponding author to researchers who provide a methodologically sound proposal. Requests made to the corresponding author (AF) will be evaluated by the Lombardy Territorial Ethics Committee
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: for another 2 years after the closure of the study
Access Criteria: request from the corresponding author approved by the Lombardy Territorial Ethics Committee

REFERENCES:
- [Result] Gavinski K, DiNardo D. Cervical Cancer Screening. Med Clin North Am. 2023 Mar;107(2):259-269. doi: 10.1016/j.mcna.2022.10.006. Epub 2022 Dec 26. PMID 36759096
- [Result] Stewart C, Ralyea C, Lockwood S. Ovarian Cancer: An Integrated Review. Semin Oncol Nurs. 2019 Apr;35(2):151-156. doi: 10.1016/j.soncn.2019.02.001. Epub 2019 Mar 11. PMID 30867104
- [Result] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer statistics, 2022. CA Cancer J Clin. 2022 Jan;72(1):7-33. doi: 10.3322/caac.21708. Epub 2022 Jan 12. PMID 35020204
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Result] Makker V, MacKay H, Ray-Coquard I, Levine DA, Westin SN, Aoki D, Oaknin A. Endometrial cancer. Nat Rev Dis Primers. 2021 Dec 9;7(1):88. doi: 10.1038/s41572-021-00324-8. PMID 34887451
- [Result] Berek JS, Matias-Guiu X, Creutzberg C, Fotopoulou C, Gaffney D, Kehoe S, Lindemann K, Mutch D, Concin N; Endometrial Cancer Staging Subcommittee, FIGO Women's Cancer Committee. FIGO staging of endometrial cancer: 2023. Int J Gynaecol Obstet. 2023 Aug;162(2):383-394. doi: 10.1002/ijgo.14923. Epub 2023 Jun 20. PMID 37337978
- [Result] Guckenberger M, Lievens Y, Bouma AB, Collette L, Dekker A, deSouza NM, Dingemans AC, Fournier B, Hurkmans C, Lecouvet FE, Meattini I, Mendez Romero A, Ricardi U, Russell NS, Schanne DH, Scorsetti M, Tombal B, Verellen D, Verfaillie C, Ost P. Characterisation and classification of oligometastatic disease: a European Society for Radiotherapy and Oncology and European Organisation for Research and Treatment of Cancer consensus recommendation. Lancet Oncol. 2020 Jan;21(1):e18-e28. doi: 10.1016/S1470-2045(19)30718-1. PMID 31908301
- [Result] Colombo N, Creutzberg C, Amant F, Bosse T, Gonzalez-Martin A, Ledermann J, Marth C, Nout R, Querleu D, Mirza MR, Sessa C; ESMO-ESGO-ESTRO Endometrial Consensus Conference Working Group. ESMO-ESGO-ESTRO Consensus Conference on Endometrial Cancer: diagnosis, treatment and follow-up. Ann Oncol. 2016 Jan;27(1):16-41. doi: 10.1093/annonc/mdv484. Epub 2015 Dec 2. PMID 26634381
- [Result] Tortorella L, Restaino S, Zannoni GF, Vizzielli G, Chiantera V, Cappuccio S, Gioe A, La Fera E, Dinoi G, Angelico G, Scambia G, Fanfani F. Substantial lymph-vascular space invasion (LVSI) as predictor of distant relapse and poor prognosis in low-risk early-stage endometrial cancer. J Gynecol Oncol. 2021 Mar;32(2):e11. doi: 10.3802/jgo.2021.32.e11. Epub 2021 Jan 11. PMID 33470061
- [Result] Ramanathan S, Tirumani SH, Ojili V. Nodal metastasis in gynecologic malignancies: Update on imaging and management. Clin Imaging. 2020 Feb;59(2):157-166. doi: 10.1016/j.clinimag.2019.11.006. Epub 2019 Nov 28. PMID 31821973
- [Result] Milam MR, Java J, Walker JL, Metzinger DS, Parker LP, Coleman RL; Gynecologic Oncology Group. Nodal metastasis risk in endometrioid endometrial cancer. Obstet Gynecol. 2012 Feb;119(2 Pt 1):286-92. doi: 10.1097/AOG.0b013e318240de51. PMID 22270280
- [Result] Fournier M, Stoeckle E, Guyon F, Brouste V, Thomas L, MacGrogan G, Floquet A. Lymph node involvement in epithelial ovarian cancer: sites and risk factors in a series of 355 patients. Int J Gynecol Cancer. 2009 Nov;19(8):1307-13. doi: 10.1111/IGC.0b013e3181b8a07c. PMID 20009882
- [Result] Woelber L, Eulenburg C, Choschzick M, Kruell A, Petersen C, Gieseking F, Jaenicke F, Mahner S. Prognostic role of lymph node metastases in vulvar cancer and implications for adjuvant treatment. Int J Gynecol Cancer. 2012 Mar;22(3):503-8. doi: 10.1097/IGC.0b013e31823eed4c. PMID 22266935
- [Result] Yang B, Zhu L, Cheng H, Li Q, Zhang Y, Zhao Y. Dosimetric comparison of intensity modulated radiotherapy and three-dimensional conformal radiotherapy in patients with gynecologic malignancies: a systematic review and meta-analysis. Radiat Oncol. 2012 Nov 23;7:197. doi: 10.1186/1748-717X-7-197. PMID 23176540
- [Result] Kidd EA, Siegel BA, Dehdashti F, Rader JS, Mutic S, Mutch DG, Powell MA, Grigsby PW. Clinical outcomes of definitive intensity-modulated radiation therapy with fluorodeoxyglucose-positron emission tomography simulation in patients with locally advanced cervical cancer. Int J Radiat Oncol Biol Phys. 2010 Jul 15;77(4):1085-91. doi: 10.1016/j.ijrobp.2009.06.041. Epub 2009 Oct 31. PMID 19880262
- [Result] Chen CC, Lin JC, Jan JS, Ho SC, Wang L. Definitive intensity-modulated radiation therapy with concurrent chemotherapy for patients with locally advanced cervical cancer. Gynecol Oncol. 2011 Jul;122(1):9-13. doi: 10.1016/j.ygyno.2011.03.034. Epub 2011 Apr 22. PMID 21514629
- [Result] Jhingran A, Winter K, Portelance L, Miller B, Salehpour M, Gaur R, Souhami L, Small W Jr, Berk L, Gaffney D. A phase II study of intensity modulated radiation therapy to the pelvis for postoperative patients with endometrial carcinoma: radiation therapy oncology group trial 0418. Int J Radiat Oncol Biol Phys. 2012 Sep 1;84(1):e23-8. doi: 10.1016/j.ijrobp.2012.02.044. Epub 2012 Apr 28. PMID 22543211
- [Result] Jereczek-Fossa BA, Ronchi S, Orecchia R. Is Stereotactic Body Radiotherapy (SBRT) in lymph node oligometastatic patients feasible and effective? Rep Pract Oncol Radiother. 2015 Nov-Dec;20(6):472-83. doi: 10.1016/j.rpor.2014.10.004. Epub 2014 Nov 7. PMID 26696788
- [Result] Ling DC, Vargo JA, Burton SA, Heron DE, Beriwal S. Salvage Curative-Intent Reirradiation Stereotactic Body Radiation Therapy for Isolated Pelvic and/or Paraortic Recurrences of Gynecologic Malignancies. Pract Radiat Oncol. 2019 Nov;9(6):418-425. doi: 10.1016/j.prro.2019.05.012. Epub 2019 May 28. PMID 31150869
- [Result] Macchia G, Lazzari R, Colombo N, Laliscia C, Capelli G, D'Agostino GR, Deodato F, Maranzano E, Ippolito E, Ronchi S, Paiar F, Scorsetti M, Cilla S, Ingargiola R, Huscher A, Cerrotta AM, Fodor A, Vicenzi L, Russo D, Borghesi S, Perrucci E, Pignata S, Aristei C, Morganti AG, Scambia G, Valentini V, Jereczek-Fossa BA, Ferrandina G. A Large, Multicenter, Retrospective Study on Efficacy and Safety of Stereotactic Body Radiotherapy (SBRT) in Oligometastatic Ovarian Cancer (MITO RT1 Study): A Collaboration of MITO, AIRO GYN, and MaNGO Groups. Oncologist. 2020 Feb;25(2):e311-e320. doi: 10.1634/theoncologist.2019-0309. Epub 2019 Oct 10. PMID 32043791
- [Result] Macchia G, Nardangeli A, Laliscia C, Fodor A, Draghini L, Gentile PC, D'Agostino GR, Balcet V, Bonome P, Ferioli M, Autorino R, Vicenzi L, Raguso A, Borghesi S, Ippolito E, Di Cataldo V, Cilla S, Perrucci E, Campitelli M, Gambacorta MA, Deodato F, Scambia G, Ferrandina G. Stereotactic body radiotherapy in oligometastatic cervical cancer (MITO-RT2/RAD study): a collaboration of MITO, AIRO GYN, and MaNGO groups. Int J Gynecol Cancer. 2022 Jun 6;32(6):732-739. doi: 10.1136/ijgc-2021-003237. PMID 35193941
- [Result] Macchia G, Pezzulla D, Campitelli M, Laliscia C, Fodor A, Bonome P, Draghini L, Ippolito E, De Sanctis V, Ferioli M, Titone F, Balcet V, Di Cataldo V, Russo D, Vicenzi L, Cossa S, Lucci S, Cilla S, Deodato F, Gambacorta MA, Scambia G, Morganti AG, Ferrandina G. Efficacy and Safety of Stereotactic Body Radiation Therapy in Oligometastatic Uterine Cancer (MITO-RT2/RAD): A Large, Real-World Study in Collaboration With Italian Association of Radiation Oncology, Multicenter Italian Trials in Ovarian Cancer, and Mario Negri Gynecologic Oncology Group Groups. Int J Radiat Oncol Biol Phys. 2023 Oct 1;117(2):321-332. doi: 10.1016/j.ijrobp.2023.04.025. Epub 2023 May 6. PMID 37150261
- [Result] Reshko LB, Baliga S, Crandley EF, Harry Lomas IV, Richardson MK, Spencer K, Bennion N, Mikdachi HE, Irvin W, Kersh CR. Stereotactic body radiation therapy (SBRT) in recurrent, persistent or oligometastatic gynecological cancers. Gynecol Oncol. 2020 Dec;159(3):611-617. doi: 10.1016/j.ygyno.2020.10.001. Epub 2020 Oct 12. PMID 33059914
- [Result] Grigsby PW, Singh AK, Siegel BA, Dehdashti F, Rader J, Zoberi I. Lymph node control in cervical cancer. Int J Radiat Oncol Biol Phys. 2004 Jul 1;59(3):706-12. doi: 10.1016/j.ijrobp.2003.12.038. PMID 15183474